CLINICAL TRIAL: NCT00145964
Title: Identification of the Genetic Variants Responsible for Primary Biliary Cirrhosis (PBC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: 04-0461-AE
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-11-29 (Estimated); Status verified 2005-08

CONDITIONS: Liver Cirrhosis, Biliary; Biliary Cirrhosis, Primary
Keywords: Biliary Cirrhosis, Primary; genes; autoimmune disease
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Primary biliary cirrhosis (PBC) is a disease of the liver, which predominantly affects women. It causes slowly progressive liver disease, which eventually causes liver failure, requiring a liver transplant. Several different studies of large patient cohorts indicate that the cause of this disease is likely due to a combination of factors including genetic and environmental. PBC is associated with several other "autoimmune diseases" - recently a gene has been identified to be abnormal in individuals with another autoimmune liver disease, namely rheumatoid arthritis. This gene usually tells the body when to switch off an immune response. This study plans to identify whether individuals diagnosed with PBC have a similar abnormality in this gene called protein Tyrosine Phosphatase.

DETAILED DESCRIPTION:
Very recently, a single nucleotide polymorphism (SNP) in the PTPN22 gene encoding the Lyp (lymphoid-specific phosphatase) PTP has been shown to be associated with susceptibility to rheumatoid arthritis (RA) and Type 1 diabetes (T1D)4,5. These data are consistent with the known role for Lyp in suppressing T cell activation and with data showing T cell activation (and potentially autoreactivity) to be increased by the RA and T1D-associated PTPN22 variant. The PTPN22 risk allele has also been recently implicated in Grave's disease and as such appears to represent a susceptibility allele for many autoimmune diseases. As a number of these conditions (RA, T1D etc.) frequently occur within members of PBC families, this PTPN22 variant is very likely to also be involved in PBC, a possibility we will directly investigate in this pilot study. The aim of this study is to analyze the frequency of a specific PTPN22 polymorphism in patients with PBC.

ELIGIBILITY:
Inclusion Criteria:

* patients attending Liver Clinic at Toronto Western Hospital, Toronto, ON, Canada
* AMA positive and liver biopsy proven PBC.

Exclusion Criteria:

- AMA negative PBC

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: E.J.L (Jenny) Heathcote, MD, Principal Investigator — UHN - Toronto Western Hospital, University of Toronto
Locations (1):
- Liver Clinic, Toronto Western Hospital, UHN., Toronto, Ontario, Canada